CLINICAL TRIAL: NCT00837603
Title: Influence of Physical Training on Cardiopulmonary Exercise Capacity and Right Ventricular Function in Patients With D-TGA and Atrial Switch Operation.
Brief Title: Physical Training in Transposition of the Great Arteries
Acronym: TrainingTGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Helmut Drexler, MD, Professor of Medicine, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TGA2009
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2011-07

CONDITIONS: Transposition of Great Vessels
Keywords: tga; atrial switch; training
MeSH Terms: conditions — Transposition of Great Vessels; DiGeorge Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training (Active Comparator): Ergometer Training
  Interventions: Behavioral: Training
- 2 (No Intervention): Counseling

INTERVENTIONS:
Behavioral: Training — Controlled home ergometer training
  Other Names: ergometer; physical exercise
  Arms: Training

SUMMARY:
In transposition patients after atrial switch operation, the morphological right ventricle serves as the systemic ventricle. These patients often develop signs of heart failure. It is not known, whether physical training can safely be recommended in these patients- like heart failure guidelines recommend training in patients with normal anatomy. Furthermore it is not known, whether these TGA-patients benefit from training with respect to cardiopulmonary exercise capacity.

DETAILED DESCRIPTION:
This is a randomized, controlled, prospective trial on the safety of physical training in TGA patients after atrial switch operation.

In transposition patients after atrial switch operation, the morphological right ventricle serves as the systemic ventricle. These patients often develop signs of heart failure. It is not known, whether physical training can safely be recommended in these patients- like heart failure guidelines recommend training in patients with normal anatomy. Furthermore it is not known, whether these TGA-patients benefit from training with respect to cardiopulmonary exercise capacity.

Primary endpoints are Systemic Ventricle Ejection Fraction and Volumes, Exercise Capacity.

Secondary endpoints are Echo Diastolic Function, as well as laboratory markers of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years

Exclusion Criteria:

* tricuspid regurgitation grade 2 or more
* sign. LVOTO or RVOTO
* pacemaker or defibrillator
* recent hospitalisation for heart failure (90 days)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Cardiac MRI Right Ventricular Ejection Fraction | 6 and 12 months
Cardiopulmonary exercise capacity | 6 and 12 months

SECONDARY OUTCOMES:
laboratory markers of heart failure | 6 and 12 months
Diastolic RV and LV function | 6 and 12 months
Right ventricular volumes | 6 and 12 months
Right ventricular mass | 6 and 12 months
NYHA-class | 6 and 12 months
quality of life questionnaire | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Roentgen, MD, Principal Investigator — Hannover Medical School; Gerd P Meyer, MD, Study Chair — Hannover Medical School; Helmut Drexler, MD, Study Director — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Westhoff-Bleck M, Schieffer B, Tegtbur U, Meyer GP, Hoy L, Schaefer A, Tallone EM, Tutarel O, Mertins R, Wilmink LM, Anker SD, Bauersachs J, Roentgen P. Aerobic training in adults after atrial switch procedure for transposition of the great arteries improves exercise capacity without impairing systemic right ventricular function. Int J Cardiol. 2013 Dec 5;170(1):24-9. doi: 10.1016/j.ijcard.2013.10.009. Epub 2013 Oct 11. PMID 24207068
- [Derived] Tutarel O, Rontgen P, Bode-Boger SM, Martens-Lobenhoffer J, Westhoff-Bleck M, Diller GP, Bauersachs J, Kielstein JT. Symmetrical dimethylarginine is superior to NT-proBNP for detecting systemic ventricular dysfunction in adults after atrial repair for transposition of the great arteries. Int J Cardiol. 2013 Oct 9;168(4):4415-6. doi: 10.1016/j.ijcard.2013.05.030. Epub 2013 May 24. No abstract available. PMID 23711443